CLINICAL TRIAL: NCT02117661
Title: ECoM Study: Effect of Carnitine Supplementation on Progression of Carotid Plaque in the Metabolic Syndrome.
Brief Title: Carnitine for the Treatment of Atherosclerosis.
Acronym: ECoM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Amer Johri (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Queen's University (Other)
Responsible Party: Sponsor-Investigator, Dr. Amer Johri, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L-Carnitine-01
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2018-11

CONDITIONS: Metabolic Syndrome
Keywords: L-carnitine; Metabolic syndrome; Atherosclerosis; Coronary artery disease; Carotid; Plaque; Cardiovascular disease; Heart disease; Vascular disease
MeSH Terms: conditions — Metabolic Syndrome; Atherosclerosis; Coronary Artery Disease; Plaque, Amyloid; Cardiovascular Diseases; Heart Diseases; Vascular Diseases | interventions — Carnitine; Cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-carnitine capsules (Experimental): 2000 mg daily (2x 500 mg capsules twice a day - BID) for six months
  Interventions: Dietary Supplement: L-carnitine capsules
- Cellulose capsules (Placebo Comparator): 2x capsules twice a day - BID (4 total per day) for six months
  Interventions: Dietary Supplement: Cellulose capsules

INTERVENTIONS:
Dietary Supplement: L-carnitine capsules — Oral
  Other Names: levocarnitine; carnitor
  Arms: L-carnitine capsules
Dietary Supplement: Cellulose capsules — oral
  Arms: Cellulose capsules

SUMMARY:
Obesity is one of the main causes of the metabolic syndrome, a condition which is becoming more common in Canada and worldwide. Metabolic syndrome is a name for a group of heart disease risk factors that occur together: obesity, diabetes, high blood pressure, and high cholesterol. These patients have a high risk of developing narrowing and blockages of blood vessels which occur when fat and cholesterol build up in the walls of blood vessels and form plaque. This is called atherosclerosis. Plaque buildup leads to stroke, heart attacks, and death. We do not understand the underlying mechanisms of the metabolic syndrome and we do not have a treatment for it. L-carnitine, a dietary supplement, has been shown to treat some components of the metabolic syndrome, but its benefit to reduce plaque in the blood vessels has never been studied. Recently there has been some controversy because a new study showed that L-carnitine could make heart disease worse in some patients. Our goal is to study whether supplementation with L-carnitine does in fact prevent or reduce buildup of plaque in blood vessels of patients with the metabolic syndrome. This novel therapy has the potential to decrease the burden of heart disease in obese and diabetic patients with the metabolic syndrome.

DETAILED DESCRIPTION:
Primary Question: Does L-carnitine (L-C) therapy slows down and/or regress atherosclerosis, as measured by total plaque volume (TPV) assessed by 3-dimensional (3D) carotid ultrasound in patients with metabolic syndrome? We hypothesize that L-C will regress atherosclerotic plaque formation.

To assess our primary outcome of L-C induced atherosclerosis regression, we anticipate a significant percent (%) difference in carotid total plaque volume (TPV) over six months of L-C treatment, compared to placebo. For our secondary outcome, we expect to show that L-C therapy compared to placebo, induces a reduction in the proportion of small-sized LDL and an increase in large LDL particles. As small dense LDL particles are more atherogenic than large buoyant ones, this would suggest a mechanism contributing to the atherosclerosis reduction induced by L-C therapy.

ELIGIBILITY:
Study Population: Patients, followed in our clinics for cardiovascular disease (CVD) prevention, fulfilling diagnosis criteria for metabolic syndrome (MetS) will be recruited. Eligibility will require a 2 step process as described.

Inclusion Criteria:

STEP 1: Initial screening; BP, weight and fasting blood samples will be obtained.

1. Men and women, >18 years, meeting the criteria for clinical diagnosis of MetS, according to the International Diabetes Federation (IDF) harmonized definition, where any 3 of the 5 following risk factors cut points constitutes a diagnosis of MetS:

   1. Elevated waist circumference: Population- and country-specific definitions; Health Canada recommends males 102 cm and women 88cm.
   2. Elevated triglycerides: 150 mg/dL (1.7 mmol/L).
   3. Reduced HDL: 40 mg/dL (1.0 mmol/L) in males; 50 mg/dL (1.3 mmol/L) in females or treated.
   4. Elevated BP: Systolic 130 and/or diastolic 85 mm Hg or treated.
   5. Elevated fasting glucose: 100 mg/dL (5.6 mmol/L), or HbA1c ≥6.2%, or treated.
2. Willing to provide informed consent. STEP 2: Baseline plaque volume ≥50 mm3 by 3D US, to ensure sufficient detectable plaque. This will be measured after consent (at Step 1), but prior to randomization/enrolment (Step 2).

Exclusion criteria:

1. Individuals who have had a change in statin and/or diabetes medication therapy or dosing in the last three months;
2. Who are actively having an unstable arrhythmia, angina or heart attack (untreated and/or unstable patients): symptomatic heart failure (NYHA 2 or greater); renal failure (GFR <50 mL/min/1.73m2);
3. Known severe abnormal blood biochemistries: Na <100 or >150 mmol/L, K <2 or >5 mmol/L, Total Serum Ca >3 mmol/L;
4. Known severe liver disease: AST >100 U/L, ALT >80 U/L, or a diagnosis of cirrhosis (Child Pugh Class A to C);
5. Known severe anemia: HgB <70 g/L;
6. Have endocrine disorders, e.g. Cushing's disease, hyper- or hypo-thyroidism;
7. Any condition expected to limit survival to less than six (6) months (ex. malignant tumor);
8. A condition limiting adherence to study procedure (i.e. alcoholism, drug addiction, known poor adherence, severe mental disorder);
9. Concomitant treatment with: anticonvulsants; L-C or derivatives; Acenocoumarol (Sintrom) and Warfarin (Coumadin) anticoagulants and vitamin K antagonists; >1g fish oil; and/or thyroid treatment;
10. A seizure disorder or at risk of seizure (CNS mass or medications that lower seizure threshold); receiving treatments for cancer or HIV infection (secondary L-C deficiency);
11. Currently pregnant or breastfeeding;
12. A history of allergy or intolerance to L-C or derivatives;
13. Vegetarians (do not eat animal flesh) due to potential for altered L-C metabolism;
14. Patients who have had a carotid surgery (ie. endarterectomy (CEA) or stent) or who are scheduled to receive carotid surgery during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Change in carotid Total Plaque Volume | Six months
  Carotid 3D ultrasound scan

SECONDARY OUTCOMES:
Change in LDL size profile | Six months
  Blood test

CONTACTS AND LOCATIONS:
Overall Officials: Amer M Johri, MD, Principal Investigator — Queen's University; J.David Spence, MD, Principal Investigator — Robarts Institute; Daren K Heyland, MD, Principal Investigator — Queen's University
Locations (2):
- Canada (2):
  - Queen's University, Cardiovascular Imaging Network at Queen's (CINQ), Kingston General Hospital, Kingston, Ontario
  - Robarts Institute, Stroke Prevention & Atherosclerosis Research Centre (SPARC), London, Ontario

REFERENCES:
- [Derived] Johri AM, Hetu MF, Heyland DK, Herr JE, Korol J, Froese S, Norman PA, Day AG, Matangi MF, Michos ED, LaHaye SA, Saunders FW, Spence JD. Progression of atherosclerosis with carnitine supplementation: a randomized controlled trial in the metabolic syndrome. Nutr Metab (Lond). 2022 Apr 2;19(1):26. doi: 10.1186/s12986-022-00661-9. PMID 35366920
- See also: Cardiovascular Imaging Network at Queen's (CINQ) — http://www.cinqlab.com